CLINICAL TRIAL: NCT05760560
Title: Incidence of Postoperative Residual Neuromuscular Blockade in the Era of Sugammadex
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Chang-Hoon Koo, Assistant professor, Seoul National University Hospital
Other Study IDs: TOF-Sugammadex
Record Dates: First submitted 2023-02-26; First posted 2023-03-08 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Postoperative Residual Curarization
MeSH Terms: conditions — Delayed Emergence from Anesthesia | interventions — Sugammadex

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Sugammadex — At the end of surgery, neuromucular blockade will be reversed with 2mg/kg or 4mg/kg sugammadex depending on the depth of neuromuscular blockade.

SUMMARY:
This study is a prospective observational study. A total 52 patients will be included in this study. We will observe the incidence of postoperative residual neuromuscular blockade in patients receiving sugammadex.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective surgery under general anesthesia.
* American Society of Anesthesiologists grade 1, 2, or 3.
* Aged >18 years

Exclusion Criteria:

* Refusal to participate in the study
* Body Mass Index < 18.5 kg/m2 or > 35 kg/m2
* History of neuromuscular disease.
* History of allergy to neuromuscular blockade
* Scheduled to transfer to the intensive care unit

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing elective surgery under general anesthesia will be screened and included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 52 (Estimated)
Dates: Start 2023-03-15 (Actual); Primary Completion 2023-08-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Postoperative residual neuromuscular blockade | On the arrival of PACU
  TOF ratio < 0.9

CONTACTS AND LOCATIONS:
Overall Officials: Chang-Hoon Koo, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Koo CH, Lee S, Yim S, Bae YK, Park I, Oh AY. Is quantitative neuromuscular monitoring mandatory after administration of the recommended dose of sugammadex? A prospective observational study. Anaesth Crit Care Pain Med. 2024 Dec;43(6):101445. doi: 10.1016/j.accpm.2024.101445. Epub 2024 Oct 16. PMID 39419348